CLINICAL TRIAL: NCT02258061
Title: Optimal Cardiac Resynchronization Therapy Pacing Rate in Non-ischemic Heart Failure Patients: a Randomized Crossover Pilot Trial.
Brief Title: Optimal Cardiac Resynchronization Therapy Pacing Rate
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Dr. Adam Ali Ghotbi, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: H-3-2011-034
Record Dates: First submitted 2014-09-29; First posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Cardiac Resynchronization Therapy; Heart Failure; Bi-ventricular Pacing; Sympathetic Activity; Quality of Life
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DDD-80 pacing (Experimental): To investigate the impact of basal pacing rates of 80-bpm (DDD-80) in CRT patients on: (i) autonomic nerve function; assessed by micro-neurography, and N-terminal pro-brain natriuretic peptide (NT-proBNP) and (ii) peak oxygen consumption (pVO2) and (iii) self-perceived quality of life (QoL).
  Interventions: Procedure: DDD-80
- DDD-60 pacing (Sham Comparator): To investigate the impact of basal pacing rates of 60-bpm (DDD-60) in CRT patients on: (i) autonomic nerve function; assessed by micro-neurography, and N-terminal pro-brain natriuretic peptide (NT-proBNP) and (ii) peak oxygen consumption (pVO2) self-perceived quality of life (QoL).
  Interventions: Procedure: DDD-60

INTERVENTIONS:
Procedure: DDD-80 — Basal pacing rate set to 80-bpm. Note:Patients have already pacemaker implanted before this study.
  Arms: DDD-80 pacing
Procedure: DDD-60 — Basal pacing rate set to 60-bpm. Note:Patients have already pacemaker implanted before this study.
  Arms: DDD-60 pacing

SUMMARY:
The optimal pacing rate during cardiac resynchronization therapy (CRT) is not known. Investigators investigate the impact of changing basal pacing frequencies on autonomic nerve function, cardiopulmonary exercise capacity and self-perceived quality of life (QoL).

DETAILED DESCRIPTION:
This is a double-blinded randomized crossover pilot study testing two basal pacing rates: DDD-60 versus DDD-80. Each patient is paced for 2 periods of 90 days with DDD-60 and DDD-80 in a randomly sequence.

Blood samples NT-proBNP plasma levels are analysed at baseline and at the end of each phase using electrochemiluminescence-immunoassay. Patients rest for 15 minutes before the samples are taken.

These result are monitored by supervisory group to ensure that increase of more than 15% than baseline values result in termination of study.

Investigators conduct two distinct questionnaires (Minnesota Living with Heart Failure (LIfHE) questionnaire and Medical Outcome Survey Short Form (SF-36)) A symptom limiting bicycle (Ergoline, Baden-Württemberg, Germany) exercise test is performed to measure maximum work capacity and oxygen consumption at each phase.

Recordings of resting muscle sympathetic nerve activity (MSNA) are sought in all patients at both rates of pacing. All patients are studied on the same set-up in the semi-recumbent position after 30 minutes of rest. Tungsten microelectrodes (Iowa Bioengineering) are inserted into the common peroneal nerve just below the knee.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with idiopathic dilated cardiomyopathy
* CRT device implanted (with initial indication in accordance with European guidelines) at least 6 months prior to inclusion.
* New York Heart Association functional (NYHA) class II-IV
* Sinus rhythm,
* Hemodynamically stable
* Biventricular pacing > 90% of the time
* On optimal medical treatment for heart failure with no changes in medications during the past 3 months.

Exclusion Criteria:

* NYHA I
* unable to perform exercise test (e.g. chronic obstructive pulmonary disease, severe arthritis)
* cancer
* plasma creatinine > 200 micromole per litre
* an admission for decompensated HF or acute coronary syndrome in the preceding 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
N-terminal pro-brain natriuretic peptide | 3 months
  Observing the change in N-terminal pro-brain natriuretic peptide in 15 patients

SECONDARY OUTCOMES:
Autonomic nerve function | 3 months
  Autonomic nerve function by micro-neurography measured in bursts/min and bursts/cardiac cycle in 15 patients
Peak oxygen consumption (pVO2) | 3 months
  pVO2 measured by a symptom limiting bicycle exercise test in 15 patients
Self-perceived quality of life | 3 months
  Measured with the LIfHE and SF-36 questionnaires in 15 patients

CONTACTS AND LOCATIONS:
Overall Officials: Adam A Ghotbi, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, University hospital of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Background] Kuniyoshi RR, Martinelli M, Negrao CE, Siqueira SF, Rondon MU, Trombetta IC, Kuniyoshi FH, Laterza MC, Nishioka SA, Costa R, Tamaki WT, Crevelari ES, Peixoto Gde L, Ramires JA, Kalil R. Effects of cardiac resynchronization therapy on muscle sympathetic nerve activity. Pacing Clin Electrophysiol. 2014 Jan;37(1):11-8. doi: 10.1111/pace.12254. Epub 2013 Aug 16. PMID 23952584
- [Background] Agostoni P, Corra U, Cattadori G, Veglia F, Battaia E, La Gioia R, Scardovi AB, Emdin M, Metra M, Sinagra G, Limongelli G, Raimondo R, Re F, Guazzi M, Belardinelli R, Parati G, Magri D, Fiorentini C, Cicoira M, Salvioni E, Giovannardi M, Mezzani A, Scrutinio D, Di Lenarda A, Mantegazza V, Ricci R, Apostolo A, Iorio A, Paolillo S, Palermo P, Contini M, Vassanelli C, Passino C, Piepoli MF; MECKI Score Research Group. Prognostic value of indeterminable anaerobic threshold in heart failure. Circ Heart Fail. 2013 Sep 1;6(5):977-87. doi: 10.1161/CIRCHEARTFAILURE.113.000471. Epub 2013 Jul 23. PMID 23881847
- [Background] Stockburger M, de Teresa E, Lamas G, Desaga M, Koenig C, Habedank D, Cobo E, Navarro X, Wiegand U. Exercise capacity and N-terminal pro-brain natriuretic peptide levels with biventricular vs. right ventricular pacing for atrioventricular block: results from the PREVENT-HF German Substudy. Europace. 2014 Jan;16(1):63-70. doi: 10.1093/europace/eut217. Epub 2013 Jul 16. PMID 23861381
- [Background] Brenyo A, Barsheshet A, Rao M, Huang DT, Zareba W, McNitt S, Hall WJ, Peterson DR, Solomon SD, Moss AJ, Goldenberg I. Brain natriuretic peptide and cardiac resynchronization therapy in patients with mildly symptomatic heart failure. Circ Heart Fail. 2013 Sep 1;6(5):998-1004. doi: 10.1161/CIRCHEARTFAILURE.112.000174. Epub 2013 Jun 25. PMID 23801020
- [Background] Shukla A, Curtis AB, Mehra MR, Albert NM, Gheorghiade M, Heywood JT, Liu Y, O'Connor CM, Reynolds D, Walsh MN, Yancy CW, Fonarow GC. Factors associated with improvement in utilization of cardiac resynchronization therapy in eligible heart failure patients: findings from IMPROVE HF. Pacing Clin Electrophysiol. 2013 Apr;36(4):433-43. doi: 10.1111/pace.12090. Epub 2013 Feb 4. PMID 23380000
- [Background] Martin DO, Day JD, Lai PY, Murphy AL, Nayak HM, Villareal RP, Weiner S, Kraus SM, Stolen KQ, Gold MR. Atrial support pacing in heart failure: results from the multicenter PEGASUS CRT trial. J Cardiovasc Electrophysiol. 2012 Dec;23(12):1317-25. doi: 10.1111/j.1540-8167.2012.02402.x. Epub 2012 Jul 25. PMID 22830441
- [Derived] Ghotbi AA, Sander M, Kober L, Philbert BT, Gustafsson F, Hagemann C, Kjaer A, Jacobsen PK. Optimal Cardiac Resynchronization Therapy Pacing Rate in Non-Ischemic Heart Failure Patients: A Randomized Crossover Pilot Trial. PLoS One. 2015 Sep 18;10(9):e0138124. doi: 10.1371/journal.pone.0138124. eCollection 2015. PMID 26382243